CLINICAL TRIAL: NCT05754775
Title: Type 2 Diabetes Remission Induced by a Korean Low-calorie Diet: A Single Center Pilot Study
Brief Title: Remission of Type 2 Diabetes Via Calorie Restriction
Acronym: K-Direct1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeouido St. Mary's Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC23ENSE0036; 2021R1A2C2013890 (Other Grant/Funding Number: the National Research Foundation of Korea)
Record Dates: First submitted 2023-02-20; First posted 2023-03-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Obesity, Morbid
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-calorie diet (Experimental): Korean low-calorie diet for type 2 diabetes
  Interventions: Behavioral: Calorie restriction via total food replacement

INTERVENTIONS:
Behavioral: Calorie restriction via total food replacement — Restricted foods designed by a clinical nutritionist that delivers to home for diabetic patients.

SUMMARY:
The primary purpose was to evaluate the efficacy of Korean low-calorie diet for obese adult patients with type 2 diabetes with a body mass index of 25 kg/m2 or higher.

DETAILED DESCRIPTION:
Previous studies reporting the natural course of type 2 diabetes generally reported progressive worsening of the disease. However, several recent studies suggested that significant weight loss induced by an very-low calorie diet could lead to the improvement in glycemic control that enough to drug discontinuation. Considering that improvement in diabetes is not permanent and hyperglycemia may recur, American and European expert groups define and express the improvement of diabetes as "remission".

In several studies in the Western contries, remission was confimed in patients who achieved significant weight loss with a daily intake of less than 800 kcal consisting of powder with high protein ingredients. When 11 patients with the disease were given only 600 kcal daily for 8 weeks, fasting blood glucose significantly decreased within 7 days. (Diabetologia 2011; 54: 2506-14). In a follow-up study, dietary intervention for 8 weeks was applied to 30 patients, about 40% of the patients showed remission of diabetes. (Diabetes Care 2016; 39: 158-65).

Based on this small study, a primary care-based research group in the United Kingdom recruited obese diabetic patients from private clinics across the country and evaluated the diabetic remission effect of a very-low caloric diet in a total of 306 patients. In this study, 46% of the intervention group and 4% of the non-intervention group reported remission, confirming a significant difference in remission rates. Patients who achieved more weight loss in the intervention group had higher remission rates, with a remission rate of 57% for patients who lost 10 to 15 kg and a remission rate of 86% for patients who lost more than 15 kg. (Lancet 2018; 391: 541-51).

On the other hand, in Korea, a study has been conducted using a Korean traditional foods designed by clinical nutritionists for diabetic patients that delivers to home. When continuous blood glucose measurement was performed while the special diet program was provided for 2 weeks, mean blood glucose and estimated glycated hemoglobin during the treatment diet period decreased compared to the free food period. The effect of the Korean-style diabetic diet was thought to be mainly due to the decrease in blood glucose levels after meals (J Korean Diabetes 2020;21:46-54).

In previous studies, total food replacement for calorie restriction was only attempted in the form of powder. In the case of the Korean diet, it contains a sufficient amount of dietary fiber and has the advantage of maintaining appropriate clinical nutrition therapy by providing various textures and tastes. Therefore, the investigators planned a clinical study to induce remission with a low-calorie diet using the Korean diet as a meal replacement therapy for calorie restriction in Korean patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes

  * If you have been diagnosed with diabetes within the last 6 years and have been treated for diabetes for more than 3 months
  * Glycated hemoglobin was measured as less than 9% without insulin treatment for the last 3 months
* Body mass index of 23kg/m2 or more

Exclusion Criteria:

* Pregnant women
* Target organ failure such as heart failure, liver failure, kidney failure, and chronic obstructive disease
* History of cardiovascular disease and cancer and current treatment
* Acute infection or acute treatment requiring hospitalization such as surgery within the last 3 months
* Any medications that may affect blood sugar within the last 6 months
* Food allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Remission | The glycated hemoglobin level in percentage measured 12 weeks after the study screening date was used.
  It is defined as a case where the HbA1c measured at the end of the 12-week intervention after stopping the drug was less than 6.5%.

SECONDARY OUTCOMES:
Weight loss | The body weight in kilograms measured 12 weeks after the study screening date was used.
  It is defined as the change in body weight before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Sang Kwon, Principal Investigator — Yeouido St. Mary's Hospital
Locations (1):
- Yeouido St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No